CLINICAL TRIAL: NCT06946836
Title: Comparison of Neoadjuvant Cadonilimab Versus Chemotherapy Combined With PD-1 in the Treatment of Resectable Non-Small Cell Lung Cancer With High PD-L1 Expression: A Single-Center, Randomized, Exploratory Clinical Study
Acronym: Neoadjuvant
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Shanghai Pulmonary Hospital, Shanghai, China, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-027
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Resectable Non-small Cell Lung Cancer; Bispecific Antibody; Neoadjuvant Therapy
Keywords: Resectable non-small cell lung cancer; bispecific antibody; Neoadjuvant therapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned in a 1:1 ratio to either the immunotherapy-combined chemotherapy group or the AK104 monotherapy group. Treatment will be administered every 3 weeks, with patients undergoing three preoperative treatment cycles before surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 monotherapy PD-1 combined with chemotherapy (Experimental): Enrolled patients will receive 3 cycles of AK104 monotherapy as neoadjuvant treatment, administered every 21 days.
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — Eligible patients will be randomly assigned in a 1:1 ratio to either the PD-1 combined with chemotherapy group or the AK104 monotherapy group. Treatment will be administered every 3 weeks, with patients undergoing three preoperative treatment cycles before surgery.
  Other Names: PD-1 combined with chemotherapy

SUMMARY:
The advent of immunotherapy has changed the treatment landscape for patients with non-small cell lung cancer. It has become the mainstay of perioperative treatment for patients with resectable non-small cell lung cancer。 Cadonilimab is the world's first bispecific antibody drug targeting PD-1 and CTLA-4. Previous studies on AK104 have demonstrated preliminary efficacy in both treatment-naïve advanced NSCLC patients and immunotherapy-resistant patients, showing a favorable safety and tolerability profile. This study aims to evaluate the effectiveness of neoadjuvant bispecific antibody AK104 compared with neoadjuvant chemotherapy combined with a PD-1 inhibitor in the treatment of resectable non-small cell lung cancer (NSCLC) with high PD-L1 expression.

DETAILED DESCRIPTION:
The advent of immunotherapy has changed the treatment landscape for patients with non-small cell lung cancer. It has become the mainstay of perioperative treatment for patients with resectable non-small cell lung cancer。 Cadonilimab is the world's first bispecific antibody drug targeting PD-1 and CTLA-4. Previous studies on AK104 have demonstrated preliminary efficacy in both treatment-naïve advanced NSCLC patients and immunotherapy-resistant patients, showing a favorable safety and tolerability profile. This study aims to evaluate the effectiveness of neoadjuvant bispecific antibody AK104 compared with neoadjuvant chemotherapy combined with a PD-1 inhibitor in the treatment of resectable non-small cell lung cancer (NSCLC) with high PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

* The patient shall sign the Informed Consent Form.

  1. Aged 18 ≥ years.
  2. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage IB-IIIA confirmed by imageological examinations (CT, PET-CT or EBUS) and Treatment-naïve for relevant antitumor therapy .
  3. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
  4. Life expectancy is at least 12 weeks.
  5. At least 1 measurable lesion according to RECIST 1.1.
  6. Patients with good function of other main organs (liver, kidney, blood system, etc.)
  7. Patients with lung function can tolerate surgery;
  8. Without systematic metastasis (including M1a, M1b and M1c);
  9. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of serplulimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
  10. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of serplulimab (whichever is later).

Exclusion Criteria:

* 1.Histology suggestive of small cell component and Participants who have received any systemic anti-cancer treatment for thymic epithelial tumor, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment and experimental treatment; 2. Participants with any unstable systemic disease (including active infection, uncontrolled hypertension), unstable angina pectoris, angina pectoris starting in the last three months, congestive heart failure (>= NYHA) Grade II), myocardial infarction (6 months before admission), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases; 3. With activate or suspectable autoimmune disease, or autoimmune paracancer syndrome requiring systemic treatment; 4. Participants who are allergic to the test drug or any auxiliary materials; 5. Participants with Interstitial lung disease currently; 6. Participants with active hepatitis B, hepatitis C or HIV; 7. Pregnant or lactating women; 8. Participants suffering from nervous system diseases or mental dieases that cannot cooperate; 9.Participated in another therapeutic clinical study; Other factors that researchers think it is not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-11 (Estimated)

PRIMARY OUTCOMES:
PCR | up to 60 months
  a complete absence of viable tumor cells in the primary tumor site and surgically removed lymph nodes after neoadjuvant treatment

SECONDARY OUTCOMES:
MPR | up to 60 months
  ≤10% residual viable tumor cells in the lung and sampled lymph nodes
ORR | up to 60 months
  a partial or complete response according to RECIST, version 1.1
OS | up to 60 months
  the time from randomization to death from any cause
EFS | up to 60 months
  the time from randomization to progression of disease, recurrence of disease, or death from any cause.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | up to 60 months
  Incidence of serious adverse events (SAEs) occurring during treatment according to NCI-CTCAE v5.0
R0 rate | up to 60 months
  Proportion of patients achieving R0 resection
Conversion rate of surgery | up to 60 months
  Conversion rate from initially unresectable to resectable NSCLC following neoadjuvant therapy

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.